CLINICAL TRIAL: NCT07015749
Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Dose of IBI3002 in Patients With Asthma - a Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: A Study to Evaluate the Safety and Tolerability of Multiple Dose of IBI3002 in Patients With Asthma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI3002T001
Record Dates: First submitted 2025-06-04; First posted 2025-06-11 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- IBI3002 600mg SC (Experimental): Participants with asthma will receive IBI3002 600mg SC
  Interventions: Drug: IBI3002
- IBI3002 150mg SC (Experimental): Participants with asthma will receive IBI3002 150mg SC
  Interventions: Drug: IBI3002
- Placebo 4ml SC (Placebo Comparator): Participants with asthma will receive Placebo 4ml SC
  Interventions: Drug: Placebo
- Placebo 1ml SC (Placebo Comparator): Participants with asthma will receive Placebo 1ml SC
  Interventions: Drug: Placebo
- Placebo 2ml SC (Placebo Comparator): Participants with asthma will receive Placebo 2ml SC
  Interventions: Drug: Placebo
- IBI3002 300mg SC (Experimental): Participants with asthma will receive IBI3002 300mg SC
  Interventions: Drug: IBI3002

INTERVENTIONS:
Drug: Placebo — Participants with asthma will receive Placebo at the corresponding dose and dosing interval.
  Arms: Placebo 1ml SC; Placebo 2ml SC; Placebo 4ml SC
Drug: IBI3002 — Participants with asthma will receive IBI3002 at the corresponding dose and dosing interval.
  Arms: IBI3002 150mg SC; IBI3002 300mg SC; IBI3002 600mg SC

SUMMARY:
This study is a randomized, double-blind, placebo-controlled study aimed at evaluating the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of IBI3002 multiple doses in participants with asthma. The study plans to enroll participants with asthma on stable inhaled treatment, FeNO≥25ppb at screening and randomization, elevated peripheral blood eosinophils and Pre-BD FEV1 ≤ 80% of the prediction. The safety, tolerability, PK, immunogenicity and changes in PD and clinical characteristics of multiple doses of IBI3002 in asthma subjects will be evaluated.

The entire study includes the screening period (4 weeks before dosing), the treatment period (12 weeks), and the safety follow-up period (8 weeks).

The study plans to enroll 9 to 27 participants with asthma, who will be randomly assigned in a 1:1:1 ratio to the following 3 cohorts to receive subcutaneous injection of the corresponding dose of IBI3002 or a matching volume of placebo. Investigators and participants will remain blind within the cohort.

Cohort 1: 150mg SC(IBI3002: placebo =2 :1); Cohort 2: 300mg SC(IBI3002: placebo =2 :1); Cohort 3: 600mg SC(IBI3002: placebo =2 :1);

The participants need to be observed at the study site for 3 hours after each dose and are allowed to leave after investigators determine no safety risk.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 65 years old (inclusive).
2. Weight ≥40kg.
3. Diagnosed with Asthma for ≥12 months in accordance with the Global Initiative for Asthma (GINA) and confirmed by the Investigator.
4. Receiving inhaled treatment with or without inhaled corticosteroids (ICS), which has been stablized for ≥ 1 month and confirmed by the Investigator.
5. FeNO ≥25ppb at screening and randomization.
6. Elevated peripheral blood eosinophils, defined as ≥300/μL in within 6 months prior to screening; OR ≥150/μL at screening.
7. Pre-bronchodilator forced expiratory volume in 1 second (pre-BD FEV) ≤ 80% of prediction.

Exclusion Criteria:

1. Co-exsiting diseases that may have an impact on the participant's own safety or participation in the study, in the opinion of the Investigator. Including but not limited to mental disorders, diseases of the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system or metabolic system.
2. A known history of active tuberculosis or clinically suspected manifestations of tuberculosis (including but not limited to pulmonary tuberculosis, lymph node tuberculosis, tuberculous pleurisy, etc.); Or chest imaging suggests the existence of suspected evidence of tuberculosis. Those with positive T-SPOT.TB need to receive preventive anti-tuberculosis treatment from 4 weeks before the first administration until the end of the study.
3. The peripheral blood white blood cells or neutrophils are lower than the lower limit of the normal value at screening or randomization.
4. Experience of life-threatening asthma attacks requiring mechanical ventilation and/or asthma attacks related to hypercapnia, respiratory failure or hypoxic epilepsy within the 5 years prior to randomization.
5. History of other lung diseases besides asthma, including but not limited to chronic obstructive pulmonary disease, interstitial lung disease, etc, in the opinion of the Investigator.

The above information is not intended to contain all considerations relevant to a participant's potential participation in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of multiple doses of IBI3002 in participants with asthma | Baseline to Week 20
  The incidence of Adverse events (AE) and Serious Adverse events (SAE) in participants with asthma after multiple administrations of IBI3002;

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic (PK) parameters of IBI3002 in participants with asthma | Baseline to Week 20
  PK parameters include, the maximum concentration (Cmax), after multiple doses.
To evaluate the pharmacokinetic (PK) parameters of IBI3002 in participants with asthma | Baseline to Week 20
  PK parameters include, the maximum concentration (Tmax), after multiple doses.
To evaluate the pharmacokinetic (PK) parameters of IBI3002 in participants with asthma | Baseline to Week 20
  PK parameters include, the maximum concentration (AUC), after multiple doses.
To evaluate the pharmacokinetic (PK) parameters of IBI3002 in participants with asthma | Baseline to Week 20
  PK parameters include the trough concentration (Cmin) after multiple doses.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China